CLINICAL TRIAL: NCT06486779
Title: A Non-interventional multiCenter Observational Study to Evaluate tHe Effectiveness and Patient-Reported Outcomes of Ofatumumab (Kesimpta®) in patieNts With Relapsing Multiple sclerOsis Treated in Routine Care Settings in Greece (CHRONOS)
Brief Title: Kesimpta (Ofatumumab) in Greek Multiple Sclerosis Patients - an Observational Study
Acronym: CHRONOS
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GGR01
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Relapsing Multiple Sclerosis (RMS)
Keywords: Relapsing Multiple Sclerosis (RMS); RMS; NIS; Greece; Ofatumumab; Kesimpta
MeSH Terms: interventions — ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- CHRONOS cohort: Patients prescribed with ofatumumab in a real world setting
  Interventions: Other: Ofatumumab

INTERVENTIONS:
Other: Ofatumumab — This is an observational study. There is no treatment allocation. The decision to initiate ofatumumab will be based solely on clinical judgement.

SUMMARY:
This study is a single-country, non-interventional, multicenter, observational study, mainly based on primary data collection to assess the effect of ofatumumab on clinical parameters of Multiple Sclerosis (MS) in a routine medical care setting, as compared to the standard of care (SoC) arm of a closely monitored phase-IIIb study (STHENOS, which includes glatiramer acetate, interferons, teriflunomide, or dimethyl fumarate)

DETAILED DESCRIPTION:
Primary data from MS adult patients who initiate ofatumumab early in their disease course will be collected over a period of two years, and will be compared to the ofatumumab and Standard of Care (SoC) arms of the STHENOS trial, a closely monitored phase-IIIb trial. Eligible patients are those with Relapsing Multiple Sclerosis (RMS) diagnosis, with 1st MS symptom within 5 years prior to ofatumumab's initiation and on treatment with ofatumumab for at least 3 months, but not longer than 6 months prior to inclusion in the study. The overall study duration is expected to be 48 months, including a recruitment period and a per-patient observation period of 24 months each. Follow-up visit frequency will be determined by the treating physician, however study-related data will be collected at study enrollment and at 6-, 12-, 18-, and 24-month data collection timepoints post with an allowable time window of ±1 month for all data collection timepoints. NEDA-3 status, MS Relapse, EDSS, MRI, PROs questionnaires, MSIS-29, SDMT, Adherence and persistence, AEs will be assessed during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written IC must be obtained before participating in the study.
2. Patients with diagnosis of RMS per McDonald Criteria (2017) and <5 years since first MS symptom prior to initiation of ofatumumab.
3. Patients who have been on treatment with ofatumumab for at least 3 months, but not longer than 6 months prior to inclusion in the study.
4. Ofatumumab treatment in line with the European Product Information of Kesimpta (i.e., adult patients with relapsing forms of MS with active disease defined by clinical or imaging features).
5. Patients with at least one available brain MRI scan performed at least 3 months after ofatumumab initiation OR for whom the physician (as per her/his routine practice and independently of his/her decision to include the patient in the current study) plans to perform such scanning within 31 days after patient's inclusion in the study.

   Notes: This MRI scan can be either brain gadolinium enhanced (Gd+) or not. In case it is not gadolinium enhanced, the most recent MRI prior to ofatumumab treatment should be brain gadolinium enhanced, for relevant comparison and identification of new lesions. This MRI scan will serve as the index reference assessment for the evaluation of NEDA-3 radiological component and shall not have been performed within 30 days after the termination of steroid therapy.
6. Patients willing and able to complete the assessments, including PRO questionnaires, as per physicians' clinical practice and as outlined in this study.

Exclusion Criteria:

1. Use of investigational drugs during the study, OR between ofatumumab initiation and inclusion into the study, OR within 3 months before ofatumumab initiation, OR within 5 half-lives of investigational drug before ofatumumab initiation, OR until the expected pharmacodynamic effect has returned to baseline, whichever is longer.
2. Currently pregnant (or intention to become pregnant within the study period), breastfeeding or lactating women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients with RMS who have initiated treatment with ofatumumab early in their disease course. Patients will have been administered ofatumumab (Kesimpta®) three to six months prior to informed consent (IC) and will continue to be treated according to the local product's prescribing information and routine medical practice in terms of visit frequency and type of assessments performed, after enrolment.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with no evidence of disease activity (NEDA-3) compared to SoC arm of STHENOS | 12 months post-enrollment for Chronos cohort and 15 months post-baseline for SoC arm of Sthenos
  Achievement of NEDA-3 status (no evidence of disease activity based on three components):
  A) No confirmed multiple sclerosis clinical relapse B) No new MRI brain activity (no new or enlarging T2 lesions, no gadolinium positive (Gd+) T1 lesions) C) No six-month confirmed disability worsening (6m-CDW).

SECONDARY OUTCOMES:
Proportion of patients achieving NEDA-3 status compared to Ofatumumab arm of STHENOS | 12 months post-enrollment for Chronos cohort and 15 months post-baseline for ofatumumab arm of Sthenos
  Achievement of NEDA-3 status (no evidence of disease activity based on three components):
  A) No confirmed multiple sclerosis clinical relapse B) No new MRI brain activity (no new or enlarging T2 lesions, no gadolinium positive (Gd+) T1 lesions) C) No six-month confirmed disability worsening (6m-CDW).
Proportion of patients achieving each individual component of NEDA-3 compared to Ofatumumab arm of STHENOS | 12 months post-enrollment for Chronos cohort and 15 months post-baseline for ofatumumab arm of Sthenos
  Achievement of NEDA-3 status and individual NEDA-3 components:
  A) Proportion of patients with no confirmed multiple sclerosis clinical relapse B) Proportion of patients with no new or enlarging T2 lesions, no gadolinium positive (Gd+) T1 lesions C) Proportion of patients with no six-month confirmed disability worsening (6m-CDW).
Proportion of patients achieving NEDA-3 status (no comparator) | 18 months post-enrollment
  Achievement of NEDA-3 status (no evidence of disease activity based on three components):
  A) No confirmed multiple sclerosis clinical relapse B) No new MRI brain activity (no new or enlarging T2 lesions, no gadolinium positive (Gd+) T1 lesions) C) No six-month confirmed disability worsening (6m-CDW).
Proportion of patients achieving each individual component of NEDA-3 (no comparator) | 18 months post-enrollment
  Achievement of NEDA-3 status and individual NEDA-3 components:
  A) Proportion of patients with no confirmed multiple sclerosis clinical relapse B) Proportion of patients with no new or enlarging T2 lesions, no gadolinium positive (Gd+) T1 lesions C) Proportion of patients with no six-month confirmed disability worsening (6m-CDW).
Proportion of patients free of 6m-RAW and 6m-PIRA - no comparator | 12 and 18 months post-enrollment
  * Proportion of patients free of 6-month confirmed relapse-associated worsening (6m-RAW)
  * Proportion of patients free of 6-month confirmed progression independent of relapse activity (6m-PIRA)
  * Proportion of patients free of both 6m-RAW and 6m-PIRA
Change in MSIS-29 impact score from enrollment. | Enrollment, 12, 18 and 24 months post-enrollment
  * Change in MSIS-29 physical impact score from enrollment.
  * Change in MSIS-29 psychological impact score from enrollment.
  The MSIS-29 is a brief self-reported measurement of the impact of multiple sclerosis on patients' quality of life (measuring 20 items for physical & 9 items for mental/psychological health), where high scores indicate worse health.
Persistence and treatment discontinuation | 24 months post-enrollment
  Proportion of patients remaining on treatment with ofatumumab and proportion of patients permanently discontinuing ofatumumab during the study.
Time from the start of ofatumumab to all-cause treatment discontinuation | 24 months post-enrollment
  Time from the start of ofatumumab to all-cause treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Greece (8):
  - Novartis Investigative Site, Alexandroupoli
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Chaïdári
  - Novartis Investigative Site, Crete Heraklion
  - Novartis Investigative Site, Ioannina
  - Novartis Investigative Site, Larissa
  - Novartis Investigative Site, Pátrai
  - Novartis Investigative Site, Thessaloniki

IPD SHARING:
Plan to Share IPD: No